CLINICAL TRIAL: NCT07342517
Title: A Phase 3 Study of NDV-01 as an Intravesical Administration to Patients With BCG-Unresponsive Non-Muscle Invasive Bladder Cancer (NMIBC), Refractory to First-line Therapy
Acronym: RESCUE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Relmada Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REL-NDV01-302
Record Dates: First submitted 2026-01-13; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer; Bladder (Urothelial, Transitional Cell) Cancer Superficial (Non-Invasive); Urothelial Carcinoma Bladder; Urothelial Carcinoma Recurrent; Urologic Cancer
MeSH Terms: conditions — Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Intervention Model Description: A Phase 3, Open-label Single-arm Study of NDV-01
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NDV-01 (sustained-release gemcitabine-docetaxel) (Experimental): Drug: NDV-01 (sustained-release gemcitabine-docetaxel) Description: Intravesical instillation of NDV-01 (sustained-release gemcitabine-docetaxel)
  Interventions: Drug: NDV-01 (sustained-release gemcitabine-docetaxel)

INTERVENTIONS:
Drug: NDV-01 (sustained-release gemcitabine-docetaxel) — Intravesical instillation of NDV-01 (sustained-release gemcitabine-docetaxel)

SUMMARY:
This is a Phase 3, open-label single-arm trial designed to evaluate the safety and efficacy of NDV-01 (sustained-release gemcitabine-docetaxel) in adult participants with NMIBC with CIS who have failed BCG therapy and who have failed first-line therapy for BCG-unresponsive NMIBC (approved or in development) and are recommended for radical cystectomy.

DETAILED DESCRIPTION:
This is a Phase 3, open-label single-arm trial designed to evaluate the safety and efficacy of NDV-01 (sustained-release gemcitabine-docetaxel) in adult participants with NMIBC with CIS who have failed BCG therapy and who have failed first-line therapy for BCG-unresponsive NMIBC (approved or in development) and are recommended for radical cystectomy.

Participants will receive an induction course and then monthly maintenance courses of NDV-1 (sustained-release gemcitabine-docetaxel) through 3 years, if there is no disease recurrence.

Participants will received an induction course of NDV-01 (6-bi-weekly intravesical instillations). Those who achieve a complete response (CR) at 3 months will be eligible for monthly maintenance instillations through year 3.

Disease status will be assessed using urine cytology, cystoscopy, and directed TURBT/biopsy (if indicated) every 3 months for the first 2 years after randomization or until disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. BCG-unresponsive NMIBC with CIS of the bladder, with or without coexisting papillary Ta/T1 tumor(s) who are ineligible for or have elected not to undergo cystectomy at the time of enrollment and have experienced 1) CIS disease within 12 months of treatment.
2. Participants with BCG-unresponsive disease must have received up to two first-line therapies or BCG-unresponsive disease and who are recommended for radical cystectomy. Such therapies may include agents approved or in development (e.g., pembrolizumab, nadofaragene firodenovec, nogapendekin alfa inbakicept-pmln, cretostimogene grenadenorepvec, detalimogene voraplasmid, TARA-002, gemcitabine intravesical system (INLEXZO®), gemcitabine, MMC, or valrubicin monotherapy. Participants will have demonstrated recurrence or intolerance after one or two first-line therapy(ies).
3. All specimens must be predominantly urothelial (transitional cell) carcinoma with or without squamous or glandular differentiation. Pure squamous or glandular tumors will not be included. Participants with less than 10% micropapillary histology will be included. All other variant histology (e.g. plasmacytoid, small cell, nested, trophoblastic variants) will not be included.

Exclusion Criteria:

1. Has had urothelial carcinoma outside of the urinary bladder (i.e., urethra, ureter, or renal pelvis) or has a predominant histological variant of UC. Ta/any T1, CIS of the upper urinary tract is allowable if treated with complete nephroureterectomy more than 24 months prior to initiating study: Participant has tumor(s) involving the prostatic urethra (ductal or stromal); N+ and/or M+ per computerized tomography (CT)/Magnetic Resonance Imagery (MR) urography. History of prior T2/T3 urothelial carcinoma of the bladder.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of NDV-01 (determined by complete response [CR] anytime) administered by intravesical instillation in patients with BCG-unresponsive NMIBC who have recurred after first-line intravesical therapy (approved or in development). | 12 months
  Percentage of participants with CR at anytime based on cystoscopy, urine cytology, and biopsies. Protocol-driven mapping biopsies (as assessed by central pathology) will be performed at 12 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein H, Teichmann R. Isotachophoretic assay of aminoglycosides and lincomycins in pharmaceuticals. J Chromatogr. 1982 Nov 26;250:152-6. doi: 10.1016/s0021-9673(00)95228-2. No abstract available. PMID 6218180
- See also: AUA/SUO Guidelines for NMIBC — https://www.auanet.org/guidelines-and-quality/guidelines/bladder-cancer-non-muscle-invasive-guideline